CLINICAL TRIAL: NCT02535065
Title: Clinical Study Plan for the Zenith® Low Profile AAA Endovascular Graft
Brief Title: Zenith® Low Profile AAA Endovascular Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Research Incorporated (Industry)
Responsible Party: Sponsor
Organization: Cook Group Incorporated (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-013 Spiral-Z
Record Dates: First submitted 2015-08-26; First posted 2015-08-28 (Estimated); Results first posted 2018-06-06 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-03

CONDITIONS: Abdominal Aortic Aneurysms; Iliac Aneurysms; Aortoiliac Aneurysms
Keywords: Low Profile; Abdominal Aortic Aneurysms; Endovascular
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Iliac Aneurysm

ARMS (1):
- Endovascular Graft (Experimental): The Zenith Low Profile AAA Endovascular Graft and ancillary components
  Interventions: Device: Zenith Low Profile AAA Endovascular Graft and ancillary components

INTERVENTIONS:
Device: Zenith Low Profile AAA Endovascular Graft and ancillary components — Treatment of patients with abdominal aortic, aortoiliac, or iliac aneurysms having morphology suitable for endovascular repair

SUMMARY:
The Zenith® Low Profile AAA Endovascular Graft Clinical Study is a clinical trial to study the safety and effectiveness of the Zenith® Low Profile AAA Endovascular Graft used in conjunction with the Zenith® Spiral-Z® AAA Iliac Leg Graft to treat abdominal aortic, aortoiliac, and iliac aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* Subject has at least one of the following

  * Aortic or aortoiliac aneurysm
  * Iliac aneurysm
  * Aneurysm with a history of growth

Exclusion Criteria:

* Less than 18 years of age
* Inability or refusal to give informed consent
* Disease considerations that would compromise patient safety or study outcomes
* Pregnant of breastfeeding or planning on becoming pregnant with 60 months
* Unwilling to comply with the follow-up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-08; Primary Completion 2017-01-23 (Actual); Study Completion 2021-01-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (37):
- United States (36):
  - Stanford University Medical Center, Stanford, California
  - University of Colorado, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - University of Florida, Gainesville, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Iowa Heart Center, West Des Moines, Iowa
  - Baptist Health Louisville, Louisville, Kentucky
  - Massachusetts General, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Borgess Research Institute, Kalamazoo, Michigan
  - Wm Beaumont Hospital, Royal Oak, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Missouri Heart Center, Columbia, Missouri
  - St. John's Mercy Medical Center, St Louis, Missouri
  - St. Vincent's Heart and Vascular Center, Billings, Montana
  - Cooper University Hospital, Camden, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - New York University - Langone Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - SUNY at Stony Brook Hospital, Stony Brook, New York
  - SUNY Upstate, Syracuse, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Summa Akron, Akron, Ohio
  - Good Samaritan-Trihealth, Cincinnati, Ohio
  - Bend Memorial Clinic, Bend, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baptist Memorial Hospital-Memphis, Memphis, Tennessee
  - Sentara Vascular Specialists, Norfolk, Virginia
  - University of Washington-Harborview Medical Center, Seattle, Washington
  - Charleston Area Medical Center, Charleston, West Virginia
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Aspirus Wausau, Wausau, Wisconsin
- Hamilton General Hospital, Hamilton, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Endovascular Graft
Started | 62
1-Month Follow-up | 62
12-Month Follow-up | 61
Completed | 42
Not Completed | 20
Not completed — Death | 13
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Arm/Group | Endovascular Graft
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.5 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 61
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 62
Diabetes [Count of Participants; unit: Participants]
  Yes | 15
  No | 47
Smoking Status [Count of Participants; unit: Participants]
  Current | 16
  Past | 40
  Never | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Without Major Adverse Events Within 30 Days
Description: Major adverse events include all-cause death, Q-wave MI, renal failure requiring dialysis, paralysis, stroke, bowel ischemia, re-intubation
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Graft
Number analyzed (Participants) | 62
Participants | 62

2. Primary Outcome: Number of Patients With Device Success
Description: Device success will be measured with none of the following: type I or III endoleaks requiring re-intervention, graft limb occlusion, aneurysm rupture or conversion to open surgical repair, aneurysm enlargement greater than 0.5 cm
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Graft
Number analyzed (Participants) | 62
Participants | 57

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Endovascular Graft
All-Cause Mortality (participants affected / at risk) | 13/62
Serious Adverse Events (participants affected / at risk) | 49/62
Other Adverse Events (participants affected / at risk) | 7/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endovascular Graft (N=62)
Angina unstable (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 6 (11)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 3 (4)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 3 (5)
Myocardial ischaemia (Cardiac disorders) | 5 (5)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (3)
Ileus (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Chest pain (General disorders) | 2 (2)
Stent-graft endoleak (General disorders) | 5 (5)
Vascular stent occlusion (General disorders) | 5 (6)
Vascular stent stenosis (General disorders) | 2 (2)
Vascular stent thrombosis (General disorders) | 1 (1)
Vessel puncture site haematoma (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (2)
Contrast media reaction (Immune system disorders) | 1 (1)
Bursitis infective (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 9 (10)
Sepsis (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Blood glucose increased (Investigations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (4)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebral small vessel ischaemic disease (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Haemorrhagic cerebellar infarction (Nervous system disorders) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Device kink (Product Issues) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hip arthroplasty (Surgical and medical procedures) | 1 (2)
Ileostomy closure (Surgical and medical procedures) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1)
Mechanical ventilation (Surgical and medical procedures) | 2 (2)
Aortic aneurysm (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Iliac artery stenosis (Vascular disorders) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endovascular Graft (N=62)
Arrhythmia (Cardiac disorders) | 4 (4)
Stent-graft endoleak (General disorders) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications from PI prior to public release and can embargo communications of trial results between 60 and 180 days from the time submitted to the sponsor for review. The sponsor can embargo publications until the sponsor has published results or 180 days has elapsed after study closure at all participating sites. The sponsor cannot restrict publication but can require changes to protect sponsor's intellectual property rights or other confidential information.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: version 6 (2013-11-06): https://cdn.clinicaltrials.gov/large-docs/65/NCT02535065/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: version 7 (2014-04-15): https://cdn.clinicaltrials.gov/large-docs/65/NCT02535065/Prot_SAP_001.pdf